CLINICAL TRIAL: NCT06817148
Title: Bicuspid Aortic Valve Replacement: EvaLuatIon of transcathetEr Versus surgEry-PILOT Trial
Acronym: BELIEVE-IT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cedars-Sinai Medical Center (Other)
Responsible Party: Principal Investigator, Raj Makkar, MD, Cedars-Sinai Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00003805
Record Dates: First submitted 2025-02-05; First posted 2025-02-10 (Actual); Last update posted 2025-02-10 (Actual); Status verified 2025-02

CONDITIONS: Aortic Valve Stenosis; Bicuspid Aortic Valve
Keywords: TAVR; BAV; SAVR
MeSH Terms: conditions — Aortic Valve Stenosis; Bicuspid Aortic Valve Disease | interventions — Transcatheter Aortic Valve Replacement

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- transcatheter aortic valve replacement (TAVR) (Active Comparator): 50% of patients will be treated with standard TAVR procedure and followed up for 10 years
  Interventions: Procedure: transcatheter aortic valve replacement (TAVR)
- surgical aortic valve replacement (SAVR) (Active Comparator): 50% of patients will be treated with standard SAVR procedure and followed up for 10 years
  Interventions: Procedure: surgical aortic valve replacement (SAVR)

INTERVENTIONS:
Procedure: transcatheter aortic valve replacement (TAVR) — percutaneous transcatheter aortic valve replacement
  Arms: transcatheter aortic valve replacement (TAVR)
Procedure: surgical aortic valve replacement (SAVR) — surgical aortic valve replacement
  Arms: surgical aortic valve replacement (SAVR)

SUMMARY:
The study protocol is a randomized trial of standard of care therapies for severe aortic stenosis (AS) in patients with a bicuspid aortic valve (BAV). Namely, the therapies to which patients will be randomized will be transcatheter aortic valve replacement (TAVR) or surgical aortic valve replacement (SAVR), in patients deemed clinically suitable for both following heart team review.

The purpose of this study is to compare the safety and efficacy of Transcatheter Aortic Valve Replacement (TAVR) versus Surgical Aortic Valve Replacement (SAVR) for treating patients with severe aortic stenosis (AS) who have a congenital bicuspid aortic valve (BAV) anatomy. Patients with BAV anatomy have been under-represented in previous trials and this study might provide important information to help guide future treatment options.

The study patients will be followed with standard of care procedures for 10 years.

ELIGIBILITY:
Inclusion Criteria:

* Provision of signed and dated informed consent form
* Stated willingness to comply with all study procedures and availability for the duration of the study
* Male or female, aged > 50 years of age
* Site-determined severe AS deemed necessary for treatment with SAVR or TAVR
* Gated contrast CT available and suitable for core laboratory analysis
* BAV anatomy confirmed by CT core laboratory analysis

Exclusion Criteria:

* Recent cardiovascular intervention within the prior 30 days.
* Presence of an existing TAVR or SAVR device
* Pregnancy or lactation
* Extreme or prohibitive TAVR or SAVR risk, determined by site or committee Active enrollment in another investigational study
* Disproportionate TAVR vs SAVR risk, as determined by treating site or committee
* Associated aortopathy (AA≥ 45 mm by maximal cross-sectional dimension, as confirmed by CT core laboratory analysis, or AA<45 mm but site plan for surgery of the aorta in the event of randomization to surgery
* Site plan for treatment of concomitant non-coronary cardiovascular disease in the event of randomization to surgery (for instance, concomitant valve surgery, septal defect or coarctation repair, aorta or root replacement or repair)
* In the presence of coronary artery disease deemed necessary for revascularization in the event of randomization to SAVR or TAVR, Syntax score ≥ 32 or deemed unsuitable for PCI, or deemed unsuitable for coronary artery bypass grafting (CABG).

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Estimated)
Dates: Start 2025-01-31 (Actual); Primary Completion 2028-02-01 (Estimated); Study Completion 2037-02-01 (Estimated)

PRIMARY OUTCOMES:
1 year hierarchical composite outcome of death, disabling stroke, non-disabling stroke, valve reintervention, rehospitalization, unfavorable KCCQ (VARC 3) | 1 year
  The primary endpoint will be analyzed by the Win ratio method14. That is, every patient in the TAVR group will be compared with every patient in the SAVR group to determine which pair has won. A win higher up in the hierarchy takes priority, so KCCQ gets used only for those pairs that were tied on the first 5 event components. Then KCCQ win is declared if the time-averaged change in KCCQ differs by 5 points or more. The win ratio= total wins on TAVR divided by total wins on SAVR, for which a 95% CI and p value is calculated.

SECONDARY OUTCOMES:
Technical success at time of exit from OR/cath lab | exit from procedure (OR or cath lab)
  defined as meeting of the following:
  * Alive
  * Successful access, delivery and retrieval of the device delivery system
  * Deployment and correct positioning (including repositioning
    /recapture if needed) of the single intended valve
  * No additional unplanned or emergency surgery or re-intervention prior to leaving OR/Cath lab related to the device or access procedure (includes need for return to bypass post initial wean
Device success | 30 days
  Defined as meeting all of the following:
  * Alive and stroke-free
  * Original intended device in place
  * No additional surgical or interventional procedures related to access or the device since completion of the original procedure (i.e., exit from the cath lab/OR)
  * Intended performance of the device:
    1. Structural performance: No migration, embolization, detachment, fracture, or thrombosis
    2. Hemodynamic performance: Mean gradient < 20mmHg, AVA >1cm2, jet velocity < 3.0 m/s
    3. Absence of the following para-device complications (PVL > mild, erosion, hemolysis, or endocarditis)
Procedural success | 30 Days
  Defined as meeting all of the following:
  1. Life-threatening bleed (BARC 3b or greater)
  2. Major vascular or cardiac structural complications requiring unplanned reintervention or surgery
  3. Stage 2 or 3 AKI (includes new dialysis)
  4. MI or need for PCI/CABG
  5. Severe heart failure or hypotension requiring IV inotrope >12 hours, ultrafiltration or mechanical circulatory support
  6. Prolonged intubation > 48 hours
  7. Need for a permanent pacemaker implant or continuous, new onset atrial fibrillation
Patient success | 1 year
  Defined as meeting all of the following:
  * Device success
  * No re-hospitalizations or re-interventions for the underlying condition (e.g., Aortic stenosis and Heart Failure)
  * Return to prior living arrangement (or equivalent)
  * Improvement in symptoms defined as increase in NYHA Class > 1 compared to Baseline
  * Improvement in functional status defined as 6MWT > 25 m compared to Baseline
  * Improvement in quality-of-life defined as KCCQ score > 10 compared to Baseline

CONTACTS AND LOCATIONS:
Overall Officials: Raj Makkar, MD, Principal Investigator — Cedars-Sinai Medical Center
Locations (1):
- Cedars-Sinai Medical Center, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No